CLINICAL TRIAL: NCT00375921
Title: Evaluation of Chemosensory Function and Taste Preference of Head and Neck Cancer Patients Prior to, On Completion of and Six Weeks After Oncology Treatment
Brief Title: Evaluating Taste and Smell Function and Food and Taste Preferences of Head and Neck Cancer Patients During Radiation Therapy/Chemotherapy
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HN-4-0028 23026
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Head and Neck Cancer
Keywords: diet; food; taste; smell; head and neck; radiation; chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Anosmia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Changes to taste and smell have been reported in head and neck cancer patients who undergo radiation and chemotherapy. This may cause food to be unappealing and can lead to a reduced food intake. Thsi study will increase our understanding of taste and smell changes and how it relates to food and taste preferences.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* diagnosed with head and neck cancer including the lip, oral cavity, salivary glands, paranasal sinuses, oropharynx, hypopharynx, larynx and thyroid
* all histologic types of cancer
* all tumour stages according to American Joint Committee for Cancer (AJCC) Staging
* all forms of RT including standard or investigational and/or concurrent standard or investigational chemotherapy for head and neck cancers
* alert and mentally competent
* English speaking

Exclusion Criteria:

* unable to swallow
* unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diagnosed with head and neck cancer including the lip, oral cavity, salivary glands, paranasal sinuses, oropharynx, hypopharynx, larynx and thyroid
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Kubrak, PhD, Principal Investigator — University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada